CLINICAL TRIAL: NCT03256409
Title: Bar and Ball Joint Overdentures Surface Roughness and Microbial Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gastrovital (Other)
Responsible Party: Principal Investigator, Valenzuela-Narváez Rocío Violeta, PhD DDS, Gastrovital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gastrovital&Development
Record Dates: First submitted 2017-07-18; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Adhesiveness
Keywords: biomaterials; methacrylates; microbiology; implant dentistry/implantology; removable prosthodontics; clinical studies/trials
MeSH Terms: interventions — Yeast, Dried

STUDY DESIGN:
Intervention Model Description: The study presents the results of a sample of ten patients randomly assigned to receive implant-retained overdentures and divided into two parallel groups of five participants in a single-blind trial at a follow-up period of 30 - 180 days permanence in the mouth. Five overdentures were made for each group: Group 1: BOD: five systems titanium bar CARES® and synOcta® Straumann® Dental Implant System, Holding AG Inc., Basel, Switzerland (BOD). Group 2: BJOD: five systems ball joint Klockner® Implant System; Soadco Inc., Escaldes-Engordany, Andorra were used in two parallel groups of five participants, in an essay to simple blind person.
Who Masked: Investigator
Masking Description: The working protocol for determining the BOD Ra and BJOD Ra and the adhesion of molds and yeasts and mesophyll aerobics was carried out entirely by an investigator and the following working methodology was considered: Information to the patient and obtainment of clinical data and patient informed consent. Patients were randomly assigned to group 1 and group 2. The saliva sample was obtained in each patient for the microbiological before the installation of the overdentures. BODs and BJODs were installed in each patient and according to each case. The BOD and BJOD were removed at 30 days for surface roughness evaluation (Ra:ųm) and the evaluation of the adhesion of mold and yeast and mesophyll aerobe (CFU/ml). For the study at 180 days the BODs and the BJODs were installed in each patient. BODs and BJODs were removed after this time to proceed to the evaluation of surface roughness and adhesion of mold and yeast and mesophyll aerobe under the same parameters mentioned above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Five Bar overdenture: BOD (Experimental): Five systems titanium bar CARES® and synOcta® Straumann® Dental Implant System, Holding AG Inc., Basel, Switzerland (Bar overdenture: Group 1) For the manufacture of the overdentures it was used as material of choice Lucitone 199® (Dentsply International Inc. York, PA) and for the adaptation of the retention systems it was used Softreliner Tough Soft® Tocuyama Dental Corporation Inc., Japan. The working protocol for determining the BOD Ra and the adhesion of molds and yeasts and mesophyll aerobics was carried out entirely by an investigator. Patients were randomly assigned to group 1. The BOD were removed at 30 - 180 days for surface roughness evaluation (Ra:ųm) and the evaluation of the adhesion of mold and yeast and mesophyll aerobe (CFU/ml).
  Interventions: Other: Adherence mold and yeast and mesophyll aerobe; Other: Surface Roughness (Ra)
- Five Ball Joint Overdenture: BJOD (Experimental): Five systems ball joint Klockner® Implant System; Soadco Inc., Escaldes-Engordany, Andorra (Ball Joint Overdenture: Group 2) For the manufacture of the overdentures it was used as material of choice Lucitone 199® (Dentsply International Inc. York, PA) and for the adaptation of the retention systems it was used Softreliner Tough Soft® Tocuyama Dental Corporation Inc., Japan. The working protocol for determining the BJOD Ra and the adhesion of molds and yeasts and mesophyll aerobics was carried out entirely by an investigator. Patients were randomly assigned to group 2. The s BJOD were removed at 30 - 180 days for surface roughness evaluation (Ra:ųm) and the evaluation of the adhesion of mold and yeast and mesophyll aerobe (CFU/ml).
  Interventions: Other: Adherence mold and yeast and mesophyll aerobe; Other: Surface Roughness (Ra)

INTERVENTIONS:
Other: Adherence mold and yeast and mesophyll aerobe — Adherence mold and yeast and mesophyll aerobe to BOD and BJOD Microbial populations have been controlled in the saliva at initial time and adherence at 30 - 180 days after the overdentures in the mouth. The saliva sample was obtained from the patient in a sterile sputum collection bottle through a sterile solution. The overdenture samples were extracted and processed for analysis. Each sample was submerged in ¼ sterile Ringer and subjected to vigorous ultrasound shaking. From each of the microbial suspensions, successive dilutions were made to determine the total number of viable microorganisms present. Total count of mold and yeast and total count of mesophyll aerobe were performed.
  Other Names: Five BOD and Five BJOD
Other: Surface Roughness (Ra) — The surface roughness of BOD and BJOD was determined with the rugosimeter the Mitutoyo Surfest SJ-301® (Mitutoyo Corporation Inc., Kanagawa, Japan), through a displacement force of 4mN and of the tray to 0.5 mm/s and back to 1 mm/s (Murtra and Arcís,1999). The roughness profile Ra was evaluated and determined in microns (ųm) through five readings for each of the samples in the study respectively.
  Other Names: Five BOD and Five BJOD

SUMMARY:
The aim of the study was to compare the surface roughness (Ra) of the implant retained mandibular bar overdenture (BOD) and the implant retained mandibular ball joint overdenture (BJOD) in jaw and its relation with the adhesion of molds and yeasts and mesophyll aerobe, in time 30 to 180 days in mouth. Five systems titanium bar CARES® and synOcta® Straumann® Dental Implant System, Holding AG Inc., Basel, Switzerland (BOD); and five systems joint ball Klockner® Implant System; Soadco Inc., Escaldes-Engordany; Andorra (BJOD), were used in two parallel groups of five participants, in an essay to simple blind person. To 30 to 180 days they were withdrawn and they were evaluated the Ra (Mitutoyo Surfest SJ-301® Mitutoyo Corporation Inc., Kanagawa, Japan) and the adhesion of microorganisms (CFU/ml).

The Ra:um (the 30th and 180th): BOD, 0.965 - 1.351; BJOD, 1.325 - 2.384. Adhesion: molds and yeasts, BOD, 2.6 x 102 and 4.6 x 103; BJOD, 3.0 x 102 and 5.3 x 104. Adhesion: mesophyll aerobe, BOD, 3.8 x 106 and 5.8 x 106; BJOD, 4.3 x 106 and 7.1 x 107. The BOD and BJOD, present different Ra (P < 0.05) to 30 to 180 days. To 30 days (P = 0.489) differences do not exist as regards the adhesion of molds and yeasts and mesophyll aerobe between both overdentures. To 180 days (P = 0.723) differences exist as regards the adhesion of mold and yeast and mesophyll aerobe, being major in BJOD.

DETAILED DESCRIPTION:
Adherence mold and yeast and mesophyll aerobe to BOD and BJOD, Surface roughness (Ra), and Statistical Analyses Microbial populations have been controlled in the saliva at initial time and adherence at 30 to 180 days after the overdentures in the mouth. The saliva sample was obtained from the patient in a sterile sputum collection bottle through a sterile solution. The overdenture samples were extracted and processed for analysis. Each sample was submerged in ¼ sterile Ringer and subjected to vigorous ultrasound shaking. From each of the microbial suspensions, successive dilutions were made to determine the total number of viable microorganisms present. Total count of mold and yeast and total count of mesophyll aerobe were performed.

The surface roughness of BOD and BJOD was determined with the rugosimeter the Mitutoyo Surfest SJ-301® (Mitutoyo Corporation Inc., Kanagawa, Japan), through a displacement force of 4mN and of the tray to 0.5 mm/s and back to 1 mm/s (Murtra and Arcís,1999). The roughness profile Ra was evaluated and determined in microns (ųm) through five readings for each of the samples in the study respectively.

The results of BOD and BJOD were compared for the determination of Ra and the adherence of mold and yeast and mesophyll aerobe. For this, we used the statistics Shapiro-Wilk, T and the Pearson Correlation Coefficient to determinate the relationship between the study variables.

ELIGIBILITY:
Inclusion Criteria:

* Total edentulous mandible from 50 to 60 years of age
* Absence of systemic conditions.

Exclusion Criteria:

* Hyperplasia and history of periodontal disease
* Patients with local and/or systemic antimicrobial treatment within 72 hours prior to evaluation during the study
* Signs of severe oral parafunction

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Average values of surface roughness (Ra) and correlation of independent test in implant-retained mandibular bar overdentures (BOD) 30 - 180 days. | Change from 30 to 180 days
  The average Ra Group 1: BOD titanium bar CARES® and synOcta Straumann® in 30 days: 0.965um. In 180 days: 1.351um. 95% confidence and Shapiro Wilk (P > 0.05), determines normal distribution. Correlation of independent test (P < 0.05) 30 days (P= 0.000) and 180 days (P=0.001) determined different Ra. Ll: Lower limit; Ul: Upper limit.
Average values of surface roughness (Ra) and correlation of independents tests in implant-retained ball joint overdentures (BJOD) 30 - 180 days. | Change from 30 to 180 days
  The average Ra Group 2: BJOD Klockner® in 30 days: 1.325um. 180 days: 2.384 um. 95% confidence and Shapiro Wilk (P > 0.05), determines normal distribution. Correlation of independent test (P < 0.05) 30 days (P=0.000) and 180 days (P=0.000) determined different Ra. Ll: Lower limit; Ul: Upper limit.

SECONDARY OUTCOMES:
Average values of mold and yeast adhesion and correlation of independents tests in implant-retained mandibular bar overdentures (BOD) and implant-retained mandibular ball joint overdentures (BJOD) 30 - 180 days | Change from 30 to 180 days
  Average adhesion values of mold and yeast. Group 1 (BOD): 30 days: 2.6 x 102 CFU/ml. Group 2 (BJOD): 30 days: 3.0 x 102 CFU/ml. Group 1 (BOD): 180 days: 4.6 x 103 CFU/ml. Group 2 (BJOD): 180 days: 5.3 x 104 CFU/ml. 95% confidence and Shapiro Wilk (P > 0.05), determines normal distribution. Correlation of independent tests 30 days (P > 0.05) BOD (P=0.051) y BJOD (P=0.052) showed no different adherence. For 180 days (P < 0.05) BOD (P=0.025) y BJOD (P=0.027) presented different adhesion. Ll: Lower limit; Ul: Upper limit
Average values of mesophyll aerobe adhesion and correlation of independents tests in implant-retained mandibular bar overdentures (BOD) and implant-retained mandibular ball joint overdentures (BJOD) 30 - 180 days | Change from 30 to 180 days
  Average adhesion values of mesophyll aerobe. Group 1 (BOD): 30 days: 3.8 x 106 CFU/ml. Group 2 (BJOD): 30 days: 4.3 x 106 CFU/ml. Group 1 (BOD): 180 days: 5.8 x 106 CFU/ml. Group 2 (BJOD): 180 days: 7.1 x 107 CFU/ml. 95% confidence and Shapiro Wilk (P > 0.05), determines normal distribution. Correlation of independent tests 30 days (P > 0.05) BOD (P=0.052) y BJOD (P=0.053) showed no different adherence. For 180 days (P < 0.05) BOD (P=0.000) y BJOD (P=0.000) presented different adhesion. Ll: Lower limit; Ul: Upper limit.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Violeta Valenzuela-Narváez, PhD DDS, Principal Investigator — CONCYTEC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stellingsma K, Slagter AP, Stegenga B, Raghoebar GM, Meijer HJ. Masticatory function in patients with an extremely resorbed mandible restored with mandibular implant-retained overdentures: comparison of three types of treatment protocols. J Oral Rehabil. 2005 Jun;32(6):403-10. doi: 10.1111/j.1365-2842.2005.01242.x. PMID 15899018
- [Result] Portmann M, Glauser R. Report of a case receiving full-arch rehabilitation in both jaws using immediate implant loading protocols: a 1-year resonance frequency analysis follow-up. Clin Implant Dent Relat Res. 2006;8(1):25-31. doi: 10.2310/j.6480.2005.00027.x. PMID 16681490
- [Result] Visser A, Meijer HJ, Raghoebar GM, Vissink A. Implant-retained mandibular overdentures versus conventional dentures: 10 years of care and aftercare. Int J Prosthodont. 2006 May-Jun;19(3):271-8. PMID 16752625
- [Result] Degidi M, Piattelli A. Immediately loaded bar-connected implants with an anodized surface inserted in the anterior mandible in a patient treated with diphosphonates for osteoporosis: a case report with a 12-month follow-up. Clin Implant Dent Relat Res. 2003;5(4):269-72. doi: 10.1111/j.1708-8208.2003.tb00210.x. PMID 15127998
- [Result] Elsyad MA, Ashmawy TM, Faramawy AG. The influence of resilient liner and clip attachments for bar-implant-retained mandibular overdentures on opposing maxillary ridge. A 5-year randomised clinical trial. J Oral Rehabil. 2014 Jan;41(1):69-77. doi: 10.1111/joor.12120. Epub 2013 Dec 20. PMID 24354686
- [Result] van Kampen F, Cune M, van der Bilt A, Bosman F. Retention and postinsertion maintenance of bar-clip, ball and magnet attachments in mandibular implant overdenture treatment: an in vivo comparison after 3 months of function. Clin Oral Implants Res. 2003 Dec;14(6):720-6. doi: 10.1046/j.0905-7161.2003.00961.x. PMID 15015948
- [Result] Lang R, Rosentritt M, Behr M, Handel G. Fracture resistance of PMMA and resin matrix composite-based interim FPD materials. Int J Prosthodont. 2003 Jul-Aug;16(4):381-4. PMID 12956492
- [Result] Panyayong W, Oshida Y, Andres CJ, Barco TM, Brown DT, Hovijitra S. Reinforcement of acrylic resins for provisional fixed restorations. Part III: effects of addition of titania and zirconia mixtures on some mechanical and physical properties. Biomed Mater Eng. 2002;12(4):353-66. PMID 12652030
- [Result] Uzun G, Keyf F. The effect of fiber reinforcement type and water storage on strength properties of a provisional fixed partial denture resin. J Biomater Appl. 2003 Apr;17(4):277-86. doi: 10.1177/0885328203017004003. PMID 12797420
- [Result] Yap AU, Mah MK, Lye CP, Loh PL. Influence of dietary simulating solvents on the hardness of provisional restorative materials. Dent Mater. 2004 May;20(4):370-6. doi: 10.1016/j.dental.2003.06.001. PMID 15019452
- [Result] Guler AU, Yilmaz F, Kulunk T, Guler E, Kurt S. Effects of different drinks on stainability of resin composite provisional restorative materials. J Prosthet Dent. 2005 Aug;94(2):118-24. doi: 10.1016/j.prosdent.2005.05.004. PMID 16046965
- [Result] Bollen CM, Lambrechts P, Quirynen M. Comparison of surface roughness of oral hard materials to the threshold surface roughness for bacterial plaque retention: a review of the literature. Dent Mater. 1997 Jul;13(4):258-69. doi: 10.1016/s0109-5641(97)80038-3. PMID 11696906
- [Result] Berger JC, Driscoll CF, Romberg E, Luo Q, Thompson G. Surface roughness of denture base acrylic resins after processing and after polishing. J Prosthodont. 2006 May-Jun;15(3):180-6. doi: 10.1111/j.1532-849X.2006.00098.x. PMID 16681500
- [Result] Keyf F, Etikan I. Evaluation of gloss changes of two denture acrylic resin materials in four different beverages. Dent Mater. 2004 Mar;20(3):244-51. doi: 10.1016/S0109-5641(03)00099-X. PMID 15209229
- [Result] Richmond R, Macfarlane TV, McCord JF. An evaluation of the surface changes in PMMA biomaterial formulations as a result of toothbrush/dentifrice abrasion. Dent Mater. 2004 Feb;20(2):124-32. doi: 10.1016/s0109-5641(03)00083-6. PMID 14706795
- [Result] Mendonca MJ, Machado AL, Giampaolo ET, Pavarina AC, Vergani CE. Weight loss and surface roughness of hard chairside reline resins after toothbrushing: influence of postpolymerization treatments. Int J Prosthodont. 2006 May-Jun;19(3):281-7. PMID 16752627
- [Result] Busscher HJ, van der Mei HC. Physico-chemical interactions in initial microbial adhesion and relevance for biofilm formation. Adv Dent Res. 1997 Apr;11(1):24-32. doi: 10.1177/08959374970110011301. PMID 9524439
- [Result] Quirynen M, Bollen CM. The influence of surface roughness and surface-free energy on supra- and subgingival plaque formation in man. A review of the literature. J Clin Periodontol. 1995 Jan;22(1):1-14. doi: 10.1111/j.1600-051x.1995.tb01765.x. PMID 7706534
- [Result] Radford DR, Challacombe SJ, Walter JD. Denture plaque and adherence of Candida albicans to denture-base materials in vivo and in vitro. Crit Rev Oral Biol Med. 1999;10(1):99-116. doi: 10.1177/10454411990100010501. PMID 10759429
- [Result] Waltimo T, Tanner J, Vallittu P, Haapasalo M. Adherence of Candida albicans to the surface of polymethylmethacrylate--E glass fiber composite used in dentures. Int J Prosthodont. 1999 Jan-Feb;12(1):83-6. PMID 10196833
- [Result] He XY, Meurman JH, Kari K, Rautemaa R, Samaranayake LP. In vitro adhesion of Candida species to denture base materials. Mycoses. 2006 Mar;49(2):80-4. doi: 10.1111/j.1439-0507.2006.01189.x. PMID 16466438
- [Result] Yildirim MS, Hasanreisoglu U, Hasirci N, Sultan N. Adherence of Candida albicans to glow-discharge modified acrylic denture base polymers. J Oral Rehabil. 2005 Jul;32(7):518-25. doi: 10.1111/j.1365-2842.2005.01454.x. PMID 15975132
- [Result] Daniluk T, Fiedoruk K, Sciepuk M, Zaremba ML, Rozkiewicz D, Cylwik-Rokicka D, Tokajuk G, Kedra BA, Anielska I, Stokowska W, Gorska M, Kedra BR. Aerobic bacteria in the oral cavity of patients with removable dentures. Adv Med Sci. 2006;51 Suppl 1:86-90. PMID 17458066
- [Result] Busscher HJ, Uyen MH, van Pelt AW, Weerkamp AH, Arends J. Kinetics of adhesion of the oral bacterium Streptococcus sanguis CH3 to polymers with different surface free energies. Appl Environ Microbiol. 1986 May;51(5):910-4. doi: 10.1128/aem.51.5.910-914.1986. PMID 3729392
- [Result] Pinna A, Zanetti S, Sechi LA, Carta F. In vitro adherence of Staphylococcus epidermidis, Serratia marcescens, and Pseudomonas aeruginosa to AcrySof intraocular lenses. J Cataract Refract Surg. 2005 Dec;31(12):2430-1. doi: 10.1016/j.jcrs.2005.08.049. No abstract available. PMID 16473245
- [Result] Shimizu K, Kobayakawa S, Tsuji A, Tochikubo T. Biofilm formation on hydrophilic intraocular lens material. Curr Eye Res. 2006 Dec;31(12):989-97. doi: 10.1080/02713680601038816. PMID 17169836
- [Result] Brusca MI, Chara O, Sterin-Borda L, Rosa AC. Influence of different orthodontic brackets on adherence of microorganisms in vitro. Angle Orthod. 2007 Mar;77(2):331-6. doi: 10.2319/0003-3219(2007)077[0331:IODOBO]2.0.CO;2. PMID 17319770
- [Result] Ryan CS, Kleinberg I. Bacteria in human mouths involved in the production and utilization of hydrogen peroxide. Arch Oral Biol. 1995 Aug;40(8):753-63. doi: 10.1016/0003-9969(95)00029-o. PMID 7487577
- [Result] Tada A, Watanabe T, Yokoe H, Hanada N, Tanzawa H. Oral bacteria influenced by the functional status of the elderly people and the type and quality of facilities for the bedridden. J Appl Microbiol. 2002;93(3):487-91. doi: 10.1046/j.1365-2672.2002.01702.x. PMID 12174048

DOCUMENTS (3):
  • Study Protocol (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT03256409/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT03256409/SAP_001.pdf
  • Informed Consent Form (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT03256409/ICF_002.pdf